CLINICAL TRIAL: NCT01871688
Title: Neuromodulation System for Pelvic Floor Dysfunction Based on the Myo-neurophysiological Assessment for Gynecological Cancer Patients
Brief Title: Pelvic Floor Rehabilitation for Gynecological Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Eun Joo Yang, Assistant professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: B-0906/077-010
Record Dates: First submitted 2013-04-16; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Female Reproductive System Neoplasm
Keywords: pelvic floor dysfunction; neuromodulation; rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- pelvic floor exercise (Other): pelvic floor rehabilitation program with neuromodulation
  Interventions: Behavioral: pelvic floor rehabilitation program with neuromodulation

INTERVENTIONS:
Behavioral: pelvic floor rehabilitation program with neuromodulation — pelvic floor rehabilitation program with neuromodulation

SUMMARY:
As cancer treatment improves, the cancer survivor's quality of life and level of function have gained increasing importance. Pelvic floor function is directly affected by gynecological cancer and treatment, and pelvic floor dysfunction (PFD) can severely affect a patient's life. PFD negatively affects health-related quality of life (HRQOL). Evaluation of PFD provides information about the disease burden and treatment-related effects directly from the patient's perspective and informs clinical decision-making. The pelvic floor musculature and sacral nerves are not easily accessible, and it is difficult to test them. Several functional assessments have been used to evaluate pelvic floor dysfunction; however, reports on methodology are sparse, and consensus on their use is lacking. Research on functional outcomes is highly complex and, consequently, must be addressed in a comprehensive framework.

DETAILED DESCRIPTION:
Patients with cervical or colorectal cancer who underwent surgery or radiotherapy are recruited for the study.

* PFM strength is measured using a perineometer (BioCon-200,McubeTechnologyCompany,Seoul,Korea). Vaginal pressure is measured using a vaginal silicon pressure sensor (cmH2O; sensitivity0.06kPa,sensitivity 5mV, threshold1.5V).
* The motor evoked potentials (MEPs) from the pelvic floor are obtained by sacral and transcranial magnetic stimulation using a Magstim 200 stimulator (Magstim Co., Whitland, Wales, UK). Patients are instructed to lie in the left lateral decubitus position,intra-anal sponge electrode (Dantec,Skovlund, Denmark)was lubricated and gently inserted into the anal canal.
* Monophasic single pulses of magnetic stimuli were delivered to the vertex corresponding to the primary motor center in the precentral gyrus using a double-cone coil(9902-00,Magstim). A figure-eight coil(9762-00,Magstim)was used to stimulate the dorsolateral area of the sacrum corresponding to the exit of the sacral cortical facilitation
* We measured the latency, amplitude, and excitability threshold(ET) of MEPs detected in pelvic floor muscles with and without facilitation. The excitability threshold at rest(RET) is defined as the lowest intensity that produced MEP responses of 100μV For optimal facilitation, we measure the latency of the MEPs with minimal contraction (10% of MVC) with RET intensity and amplitude with a moderate contraction
* Patient-reported HRQOL Quality of life General and condition-specific aspects of HRQOL were assessed using the EORTC QLQ-C30 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women with gynecological cancer who had radical hysterectomy and pelvic lymph node dissection

Exclusion Criteria:

* infectious diseases of the urinary tract and vagina

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Amplitude (uV) of motor evoked potential (MEP) evoked by magnetic stimulation on the sacral plexus. | 1week after intervention
  We measure the amplitude (uV) of motor evoked potential (MEP) evoked by magnetic stimulation on the sacral plexus at the baseline and 1wk after intervention. Then we compare the change of the amplitude (1 wk after intervention-baseline)between two groups.

SECONDARY OUTCOMES:
pelvic floor muscle strength(mmHg) | baseline, up to 1week after intervention
  We measure the pelvic floor muscle strength using perometer (mmHg)at baseline and 1 wk after intervention then compare the change of pelvic floor muscle strength(1wk after intervention-baseline) between two groups.
latency (ms) of MEP (motor evoked potential) | baseline, up to 1week after intervention
  We measure the latency (ms) of MEP evoked by magnetic stimulation on the sacral plexus and compare the change of latency (1wk after intervention-baseline)between two groups
Functional score and symptom scale of QuEORTC QLQ-C-30,EORTC CX-24 | baseline, up to 1week after intervention
  We evaluate the functional score and symptom scale with EORTC QLQ-C30, EORTC QLQ-CX24 questionnaires and compare the change between two groups.
Total Bladder, bowel,sexual functional scores measured by the pelvic floor questionnaire | baseline, up to 1week after intervention
  We evaluated the bladder, bowel, sexual functional scores with the interviewer-administered pelvic floor questionnaire at baseline and 1wk after intervention then compare the change of the scores between two groups
Hiatal dimension (mm) and levator plate angle (º) on maximal pelvic floor muscle contraction measure with ultrasound | baseline, up to 1week after intervention
  We measure the Hiatal dimension (mm) and levator plate angle (º) on maximal pelvic floor muscle contraction using ultrasound with curved transducer (3.5-6 MHz)at baseline and 1 wk after intervention and compare the change between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Eun Joo Yang, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea